CLINICAL TRIAL: NCT00986531
Title: A Single Center, Double-Blind, Randomized, Placebo-Controlled, Two-Period Crossover Study to Access an Early Signal of Efficacy for Cognition and Negative Symptoms With AZD8529 in Patients With Schizophrenia
Brief Title: The Effects AZD8529 on Cognition and Negative Symptoms in Schizophrenics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D2285M00016
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Schizophrenia
Keywords: schizophrenia; early phase trials
MeSH Terms: conditions — Schizophrenia | interventions — AZD8529

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): 80 mg AZD8529
  Interventions: Drug: AZD8529
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo to match AZD8529

INTERVENTIONS:
Drug: AZD8529 — 2 capsules by mouth for 3 days
  Arms: 1
Drug: Placebo to match AZD8529 — 2 capsules by mouth for 3 days
  Arms: 2

SUMMARY:
The purpose of this study is to assess if AZD8529 improves performance on neurobehavioral probes of attention, working memory and affective reactivity in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizoaffective disorder

Exclusion Criteria:

* ECT in the last 6 months
* Substance abuse or dependence
* History of claustrophobia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2009-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) | 1 fMRI on Day 4; 1 fMRI on Day 21
Computerized neurocognitive tests | 1 on Day -1; 1 on Day 1 and on Day 21

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Day-1; Day 4; Day 17; Day 21
Electroencephalography (EEG) | Day 4; Day 21
Laboratory assessment: electrocardiogram (ECG), physical exam, vital signs, | Labs at screening and on Days -1, 4, 17, 21, and 35; ECG at screening and Day 35; Physical Exam at screening and Day 35; Vital signs at screening and Days -1,4, 17, 21, and 35
Suicidality assessment, collection of adverse events | Suicidality assesment at screening; and Days -1, 4, 17, 21, and 35 Adverse events at screening, and Days -1,4,17,21, and 35

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Gur, Principal Investigator — Hospital of the University of Pennsylvania, Dept of Psychiatry, Neuropsychiatry Section
Locations (1):
- Research Site, Philadelphia, Pennsylvania, United States